CLINICAL TRIAL: NCT05741359
Title: A Phase I/II Clinical Study of the Safety and Efficacy of CD19-targeted Non-viral PD1 Site-specific Integrated CAR-T Cell Injection (BRL-201) in the Treatment of Relapsed or Refractory B Lymphocyte Non-Hodgkin Lymphoma
Brief Title: The Safety and Efficacy of BRL-201 in the Treatment of r/r B Lymphocyte Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bioray Laboratories (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other); Zhejiang University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-BRL-201
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Non-hodgkin Lymphoma,B Cell

STUDY DESIGN:
Intervention Model Description: Total target count of CD3+CAR+ viable cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): 5- 10.0×10^6/kgBW
  Interventions: Drug: CD19-targeted non-viral PD1 site-specific integrated CAR-T cell injection

INTERVENTIONS:
Drug: CD19-targeted non-viral PD1 site-specific integrated CAR-T cell injection — CD19-targeted non-viral PD1 site-specific integrated CAR-T cell injection
  Other Names: BRL-201

SUMMARY:
This is a multi-center, single-arm, open-label clinical study, and the sample size is set to 12-18 subjects.

DETAILED DESCRIPTION:
This is a multi-center, single-arm, open-label clinical study, and the sample size is set to 12-18 subjects. Based on the "3 + 3" dose escalation design principle, subjects will be divided into 3 groups from low dose to high dose in sequence (Group A; Group B; Group C. Additional subjects will be enrolled into the RP2D group to ensure that 6-9 efficacy-evaluable subjects are available in the RP2D group before entering the phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in this clinical study and sign an informed consent form;
2. Age ≥ 18 years old;
3. Estimated survival time ≥ 3 months;
4. Presence of at least one measurable lesion as assessed according to Lugano Classification 2014 for response assessment in lymphomas (i.e., the cross-sectional images obtained by CT show that the long diameter of lymph node lesions is > 15 mm or the long diameter of extranodal lesions is > 10 mm, and FDG-PET scan results are positive). Lesions, for which radiotherapy was provided, can be regarded as measurable lesions only if there is an unequivocal progression after radiotherapy;
5. Histopathologically confirmed aggressive B-NHL; positive expression of CD19 in tumors detected by immunohistochemistry or flow cytometry; pathological types of B-NHL (according to WHO Lymphoma Classification 2016);
6. Relapsed or refractory diseases;
7. Subjects who must receive adequate prior therapy;
8. Absence of invasion of central nervous system (CNS) lymphoma by cranial magnetic resonance imaging (MRI);
9. Hematological parameters meeting the requirements;
10. Blood biochemistry meeting the requirements;
11. LVEF ≥ 55%;
12. No severe pulmonary disorders;
13. Toxic reactions induced by prior anti-lymphoma therapy must be stable and resolved to grade ≤ 1;
14. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
15. Patients with physical conditions for apheresis of peripheral blood; 16 . Willing to abide by the rules formulated in the study protocol.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Subjects who previously received allogeneic cell therapies, including allogeneic stem cell transplant;
3. Subjects who previously received anti-CD19 targeted therapy, except those who receive BRL-201 and are eligible to receive reinfusion in this study;
4. Prior treatment with any CAR-T cell product or other genetically modified T cell therapies;
5. History of Richter's transformation of chronic lymphocytic leukemia (CLL);
6. Presence of uncontrollable fungal, bacterial, viral, or other infections requiring systemic therapy. Patients can be enrolled if the simple urinary tract infection or pharyngitis responds to treatment;
7. Subjects with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood HBV DNA titer higher than the upper limit of detection; hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; human immunodeficiency virus (HIV) antibody positive; syphilis test positive;
8. Severe mental disorders; history of CNS disorders (e.g., epileptic seizure, cerebrovascular ischemia/hemorrhage, dementia, cerebellar diseases, or any CNS-involved autoimmune disorders);
9. Active autoimmune disorders requiring immunotherapy, including but not limited to end organ damages caused by autoimmune disorders (e.g., Crohn's disease, rheumatoid arthritis, and systemic lupus erythematosus) in the past 2 years, or requiring systemic application of immunosuppressive drugs or other drugs for systemic control of diseases;
10. Primary immunodeficiency;
11. History of other malignancies;
12. Patients with severe cardiovascular disorders, including but not limited to those with lymphoma infiltration in the cardiac atrium or ventricles and those with a history of myocardial infarction, cardioangioplasty or stent implantation, unstable angina, or other clinically significant heart diseases within 12 months before enrollment;
13. History of deep venous thrombosis or pulmonary embolism within 6 months before enrollment;
14. Patients who are receiving oral anticoagulant therapy; prothrombin time (PT), activated partial thromboplastin time (APTT), or international normalized ratio (INR) > 1.5 × ULN without anticoagulant therapy;
15. Presence of any indwelling tube or catheter (e.g., tube or catheter for percutaneous nephrostomy, indwelling catheter, or catheter in pleural cavity/peritoneal cavity/pericardium). Dedicated central venous access catheters (e.g., Port-a-Cath or Hickman catheter) are permitted;
16. Lymphoma cells detected in cerebrospinal fluid, presence of brain metastases, history of CNS lymphoma, or history of lymphoma cells detected in cerebrospinal fluid or brain metastases;
17. Conditions (e.g., intestinal obstruction or vascular compression) requiring emergency treatment due to tumor masses;
18. History of severe immediate hypersensitivity to any drug to be used in this study;
19. Vaccination of live vaccines, excluding corona virus disease 2019 (COVID-19) vaccines, within ≤ 6 weeks before the start of the pretreatment regimen;
20. Any circumstances that possibly increase the risk of subjects or interfere with the study results as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
DLT | Within 28 Days After BRL-201 Infusion
  The number and severity of dose-limiting toxicity (DLT) events
AEs | Up to 24 Months After BRL-201 Infusion
  The total number, incidence, and severity of AEs
RP2D | Within 28 Days After BRL-201 Infusion
  The recommended phase 2 dose

CONTACTS AND LOCATIONS:
Overall Officials: Wei Li, Study Chair — Bioray Laboratories
Locations (3):
- China (3):
  - Wuhan Union Hospital, Wuhan, Hubei
  - Tianjin Institute of Hematology, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No